CLINICAL TRIAL: NCT07396272
Title: A Pilot, Open-label Phase II Trial of Adjunctive Treatment With Ketamine Hydrochloride Prolonged-Release Tablets (KET01) During the Initiation of Antidepressant Therapy in Major Depressive Disorder
Brief Title: A Clinical Trial of Add-on Oral Slow-release Ketamine Treatment in Major Depression
Acronym: KET01-IIT03
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel Lindqvist (Other)
Collaborators: Ketabon (Unknown); Lund University (Other)
Responsible Party: Sponsor-Investigator, Daniel Lindqvist, Head of Psychiatry Division and research, Principal Investigator, Senior Consultant, Region Skane
Organization: Region Skane (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-524841-28-00
Record Dates: First submitted 2025-12-15; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine-treated (Experimental): Only arm of this pilot study, all 12 patients enrolled will be included in this arm. Treated with Ketamine Hydrochloride Prolonged-Release Tablets (KET01, 240 mg) for one week (8 days) with four doses.
  Interventions: Drug: Treatment with Ketamine Hydrochloride Prolonged-Release Tablets

INTERVENTIONS:
Drug: Treatment with Ketamine Hydrochloride Prolonged-Release Tablets — Only intervention of this pilot study, administered to all 12 patients enrolled. Treatment with Ketamine Hydrochloride Prolonged-Release Tablets (KET01, 240 mg) for one week (8 days) with four doses.

SUMMARY:
* The goal of this clinical trial is to explore if the treatment with ketamine tablets in addition to standard antidepressant therapy can reduce depressive symptoms in adults with Major Depressive Disorder. The main question it aims to answer is: Does adjunctive ketamine therapy reduce depressive symptoms after one week of treatment compared to baseline, measured by the Montgomery-Åsberg Depression Rating Scale (MADRS)?
* Participants will start ketamine treatment together with a new standard antidepressant. During the treatment week, patients will receive four doses of Ketamine Hydrochloride Prolonged-Release Tablets (240 mg) at the clinic. They will fill in different questionnaires and rating scales during screening, treatment and follow-up, and will leave blood samples at five of the visits to monitor side effects and identify possible biomarkers. After a week, the ketamine treatment is finished while the standard antidepressant therapy continues. The participation in this trial is completed after three aditional weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given their written consent to participate in the trial.
* BMI ≥ 18 and ≤ 35 kg/m2.
* Primary diagnosis of MDD meeting DSM-5-TR criteria and one of the following episode characteristics: (a)MDD, single episode, moderate (ICD-10-CM: F32.1); (b) MDD, single episode, severe, without psychotic features (ICD-10-CM: F32.2); (c) MDD, recurrent, moderate (ICD-10-CM: F33.1); (d) MDD, recurrent, severe, without psychotic features (ICD-10-CM: F33.2)
* Duration of current depressive episode no longer than 12 months prior to screening.
* MADRS score ≥ 22 at screening
* Willingness to start a new, conventional antidepressant treatment which is chosen by the treating physician with regards to side effect profile and previous treatments, together with KET01, dosed according to the prescribed schedule.
* Willingness to terminate any ongoing antidepressant treatment if deemed ineffective by study physician in accordance with clinical practice (tapering or immediate stop), followed by a wash-out phase of at least 7 days without medication before treatment with the new antidepressant is initiated together with KET01.
* For females of childbearing potential: Must be willing to undergo pregnancy tests and will be required to use highly effective contraceptive measures from the time of informed consent until 28 days after last IMP intake. Methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral or injectable); implantable intrauterine device (IUD); intrauterine hormone-releasing system (IUS), bilateral tubal occlusion or practicing sexual abstinence (if this is in line with the preferred and usual lifestyle of the participant).
* For male participants with a partner of childbearing potential: Must be willing to use adequate contraceptive measures (barrier method) or practice sexual abstinence (if this is in line with the preferred and usual lifestyle of the participant) from the time of informed consent until 28 days after last IMP intake. Note: These requirements also apply for male participants who have had a vasectomy.

Exclusion Criteria:

* Known hypersensitivity or intolerance to ketamine or any of the excipients.
* Pregnancy, breastfeeding or planned pregnancy (if female).
* High suicide risk according to the overall assessment of the research physician.
* Known psychiatric and neurological concomitant condition of:

MDD, single episode, severe, with psychotic features (ICD-10-CM: F32.3), MDD, recurrent, severe, with psychotic features (ICD-10-CM: F33.3), Schizophrenia spectrum and other psychotic disorders (ICD-10-CM: F21, F22, F23, F20.81, F20.9, F25.0, F25.1, F06.0, F06.1, F06.2, F28 and F29) or bipolar disorder (ICD-10-CM: F31), other mental disorder due to known physiological condition (ICD-10-CM: F06). Participants with first-degree relatives (parents, brothers, sisters or children) with psychotic or bipolar disorders are also not considered eligible. Paranoid or schizoid personality disorder (ICD-10-CM: F60.0, F60.1). Antisocial, borderline, histrionic or narcissistic personality disorder (ICD-10-CM: F60.2, F60.3, F60.4, F60.81). Neurodevelopmental disorders, e.g. moderate to profound intellectual developmental disorders (ICD-10-CM: F71, F72, F73), or autism spectrum disorders (ICD-10-CM: F84).

* Known or suspected lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder, epilepsy (excluding uncomplicated childhood febrile seizures with no sequelae) or any other disease/procedure/accident/intervention which, according to the investigator is deemed associated with significant injury to or malfunction of the CNS.
* History of significant head trauma within the past 2 years prior to Visit 1.
* History of cerebrovascular event (e.g. stroke, prolonged ischaemic neurologic deficit [PRIND], transient ischaemic attack).
* Known or suspected ongoing cardiac disease (e.g. unstable angina, congestive heart failure, tachyarrhythmia or myocardial infarction).
* Clinically significant abnormal electrocardiogram findings at Visit 1 which may jeopardize participant's safety according to the investigator.
* Untreated or uncontrolled hypertension (after 5 minutes of rest, systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 120 mmHg confirmed by three sequential measurements with at least 5 minutes between the single measurements).
* Laboratory findings suggesting impaired hepatic function or liver cirrhosis i.e. gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values > 2x times the upper limit of normal (ULN) or total bilirubin > 1.5 times the ULN at Visit 1. Participants with an isolated increase of indirect bilirubin not previously documented as a diagnosis of Gilbert's syndrome must be discussed with the medical monitor.
* Known hepatitis B or C.
* eGFR < 60 mL/min/1.73 m2 or creatinine > 200 μmol/L at Visit 1 or ongoing dialysis or kidney transplants.
* Diabetes mellitus with a haemoglobin A1c (HbA1c) value > 64 mmol/mol at the screening visit.
* Hyperthyroidism.
* Uncontrolled hypothyroidism i.e. not at stable treatment with thyroid hormones (triiodothyronine/thyroxine [T3/T4]) within the 6 weeks before Visit 1 or abnormal thyroid stimulating hormone (TSH) and free thyroxine (fT4) values at Visit 1.
* History (within 5 years before Visit 1) of complicated cystitis (defined as cystitis in males; due to anatomical abnormalities; due to immunocompromised state, in pregnant women; recurrent infections despite adequate treatment; infections occurring after instrumentation such as nephrostomy).
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the trial, or jeopardise the conduct of the trial according to the protocol.
* Previous administration of ketamine (with exception of known or suspected ketamine-anaesthesia) or esketamine.
* Prohibited prior and concomitant therapies and medication (see 7.3 Concomitant use of other medicinal products and treatments).
* History of moderate to severe alcohol use disorder or substance use disorder, including e.g. benzodiazepines, opiates, ketamine, hallucinogens and related drugs, stimulants (e.g. phencyclidine [PCP]), lysergic acid diethylamide [LSD], 3,4-methylenedioxymethamphetamine [MDMA], dextromethorphan, amphetamines, cocaine) or cannabis, except nicotine and caffeine, within 6 months before Visit 1 or a positive drug abuse test except for allowed medication prescribed for a medical condition.
* Participation in other treatment studies.
* Ongoing electroconvulsive treatment (ECT) or repetitive transcranial magnetic stimulation (rTMS).
* Ongoing compulsory psychiatric care.
* Other reason, as assessed by the investigator, that prevents the research subject's participation such as risk that the subject is unable to complete the trial (non-compliance).
* Recently started psychotherapy (within 6 weeks) or planning to start such treatment during participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) after one week of treatment compared to baseline visit | Between day 1 (baseline visit) and day 8 (day of last dosing)
  * In MADRS, 10 items are rated with a score of 0 to 6 (total score: 0 to 60). A higher MADRS score indicates more severe depression.
  * Cut-off points: 0 to 6: normal/symptom-free, 7 to 19: mild depression, 20 to 34: moderate depression 35 to 60: severe depression.

SECONDARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score at other timepoints than the primary endpoint | Between day 1 (baseline visit) and visits on day 3, 5, 15 and 29
  * In MADRS, 10 items are rated with a score of 0 to 6 (total score: 0 to 60). A higher MADRS score indicates more severe depression.
  * Cut-off points: 0 to 6: normal/symptom-free, 7 to 19: mild depression, 20 to 34: moderate depression 35 to 60: severe depression.
Change in Clinical Global Impression - Severity (CGI-S) rating scale from baseline to every post-baseline measurement (day 3, 5, 8, 15, 29) | Between day 1 (baseline visit) and visits on day 3, 5, 15 and 29
  In CGI-S, the overall illness severity is rated from 1 to 7:
  * 1: Normal, not at all ill
  * 2: Borderline mentally ill
  * 3: Mildly ill
  * 4: Moderately ill
  * 5: Markedly ill
  * 6: Severely ill
  * 7: Among the most extremely ill patients
Total score of Clinical Global Impression - Efficacy Index (CGI-E) rating scale at every post-baseline measurement (day 3, 5, 8, 15, 29) | Between first evaluation after treatment start (day 3) and last follow-up visit (day 29)
  The CGI-E is rated using a 4 × 4 matrix, consisting of:
  Therapeutic Effect:
  1 = Marked; 2 = Moderate; 3 = Minimal; 4 = None
  Side Effects:
  1 = None; 2 = Do not significantly interfere with functioning; 3 = Significantly interfere with functioning; 4 = Overwhelming and intolerable The CGI-E result is recorded as a paired score (e.g., 2:1, indicating a moderate therapeutic effect with no adverse effects). Investigators should base their evaluation on all available clinical information, including observed symptom changes, participant-reported outcomes, and the nature and impact of any adverse events.
Change in Patient Health Questionnaire-9 (PHQ-9) and the composite inflammatory depressive symptom score (InfDep score) consisting of PHQ-9 items # 3, 4 and 5 between baseline (day 1) and the two follow-up visits (day 15 and 29) | Between baseline visit (day 1) and last follow-up visit (day 29)
  In PHQ-9, 9 items are rated with a score of 0 to 3 from being experienced never (0) to almost every day (3) during the last 2 weeks (total score: 0 to 27). A higher PHQ-9 score indicates more severe depression. Cut-off points: 0-4: None to minimal depression, 5-9: Mild depression, 10-14: Moderate depression, 15-19: Moderately severe depression, 20-27: Severe depression
Change in generalized anxiety disorder-7 (GAD-7) between baseline (day 1) and two follow-up visits (day 15 and 29) | Between baseline visit (day 1) and last follow-up visit (day 29)
  In GAD-7, 7 items are rated with a score of 0 to 3 from being experienced never (0) to almost every day (3) during the last 2 weeks (total score: 0 to 27). A higher GAD-7 score indicates more severe anxiety. Cut-off points: 0-4: No to low anxiety, 5-9: Mild anxiety, 10-14 Moderate anxiety, 15+ Severe anxiety.
Change in Columbia Suicide Severity Rating Scale (C-SSRS) between baseline and three post-baseline visit (day 8, 15, 29) | Between baseline visit (day 1) and last follow-up visit (day 29)
  In C-SSRS, suicidality is mapped by yes/no questions and rating scales from 1 to 5. The higher the score on these scales, the more severe is the suicidality.
Response rate (≥ 50% decrease from baseline in MADRS total score) at every post-baseline visit (day 3, 5, 8, 15, 29). | Between first evaluation after treatment start (day 3) and last follow-up visit (day 29)
  * In MADRS, 10 items are rated with a score of 0 to 6 (total score: 0 to 60). A higher MADRS score indicates more severe depression.
  * Cut-off points: 0 to 6: normal/symptom-free, 7 to 19: mild depression, 20 to 34: moderate depression 35 to 60: severe depression.
Remission rate (MADRS score of ≤10) at every post-baseline visit (day 3, 5, 8, 15, 29). | Between first evaluation after treatment start (day 3) and last follow-up visit (day 29)
  * In MADRS, 10 items are rated with a score of 0 to 6 (total score: 0 to 60). A higher MADRS score indicates more severe depression.
  * Cut-off points: 0 to 6: normal/symptom-free, 7 to 19: mild depression, 20 to 34: moderate depression 35 to 60: severe depression.
Change in sedentary behaviour (SED) between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of determining physical activity measured by wearable activity meters
Change in light physical activity (LPA) between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of determining physical activity measured by wearable activity meters
Change in moderate- to vigorous physical activity (MVPA) between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of determining physical activity measured by wearable activity meters
Change in number of steps between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of determining physical activity measured by wearable activity meters
Change in total sleep time (TST) between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of analysing changes in sleep pattern measured by wearable activity meters
Change in sleep efficiency (SE) between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of analysing changes in sleep pattern measured by wearable activity meters
Change in wake after sleep onset (WASO) between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of analysing changes in sleep pattern measured by wearable activity meters
Change in number of awakenings (NA) between baseline (day 1) and every post-baseline visit (day 3, 5, 8, 15, 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Parameter is part of analysing changes in sleep pattern measured by wearable activity meters
Concentration of the inflammatory biomarker high-sensitive C-reactive protein in the blood plasma at baseline (day 1) and three post-baseline visits (day 8, 15, 29) | Between baseline visit (day 1) and last follow-up visit (day 29).
Concentration of the inflammatory biomarker interleukin-6 in the blood plasma at baseline (day 1) and three post-baseline visits (day 8, 15, 29) | Between baseline visit (day 1) and last follow-up visit (day 29).
Concentration of the inflammatory biomarker tumor necrosis factor alpha in the blood plasma at baseline (day 1) and three post-baseline visits (day 8, 15, 29) | Between baseline visit (day 1) and last follow-up visit (day 29).
Concentration of the inflammatory biomarker white blood cell count in the blood plasma at baseline (day 1) and three post-baseline visits (day 8, 15, 29) | Between baseline visit (day 1) and last follow-up visit (day 29).
Change in Connor-Davidsson Resilience Scale (CD-RISC-25) between baseline (day 1) and two post-baseline visits (day 8 and 29) | Between baseline visit (day 1) and last follow-up visit (day 29)
  In CD-RISC-25, 25 statements are rated with a score of 0 to 4 from being not true at all (0) to true almost all the time (4) (total score: 0 to 100). A higher CD-RISC-25 score indicates higher resilience.
Change in genomic DNA methylation patterns between baseline and two post-baseline visits (day 8 and day 29). | Between baseline visit (day 1) and last follow-up visit (day 29)
  Genomic DNA for DNA methylation analysis will be purified from whole blood using a commercially available kit. DNA methylation will be assessed using the Infinium MethylationEPIC v2.0 BeadChip array, covering > 900 000 unique methylation sites. Quality metrics will include assessment of bisulfite conversion efficiency using built-in control probes, evaluation of overall signal intensities across samples, and identification of outlier samples through inspection of quality control (multidimensional scaling) plots. Probes will be filtered to remove those with detection p-value >0.01 in >5% of samples, probes with known single nucleotide polymorphisms (SNPs) at the CpG interrogation site or single base extension site, cross-reactive probes that map to multiple genomic locations. For differential methylation analysis, β-values will be transformed to M values using logit transformation to stabilise variance and approximate normality.
Patient's personal experience with effect of ketamine treatment on mood | At the last follow-up (day 29)
  Qualitative interview with open-ended question

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lindqvist, PhD, MD, Principal Investigator — Region Skåne
Locations (1):
- Adult Psychiatry, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No